CLINICAL TRIAL: NCT05130268
Title: Pragmatic Randomized Clinical Trial of Early Dronedarone Versus Usual Care to Change and Improve Outcomes in Persons With First-Detected Atrial Fibrillation
Brief Title: Early Dronedarone Versus Usual Care to Improve Outcomes in Persons With Newly Diagnosed Atrial Fibrillation
Acronym: CHANGE-AFIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Heart Association (Other)
Collaborators: Duke Clinical Research Institute (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 176131-M
Record Dates: First submitted 2021-10-27; First posted 2021-11-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Arrhythmias, Cardiac; Atrial Fibrillation; Anti-Arrhythmic Agents; Heterocyclic Compounds; Dronedarone; Multaq
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Dronedarone

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, open-label, pragmatic clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronedarone (Experimental): In most patients, the investigators anticipate usual care to include an atrioventricular nodal blocking agent (beta-blocker, non-dihydropyridine calcium channel blocker, or digoxin) without an antiarrhythmic. As dronedarone has anti-adrenergic rate controlling properties, a low dose of beta-blocker or calcium-channel blocker is recommended in the United States Prescribing Information (USPI) when starting dronedarone. In the dronedarone arm concomitant digoxin use will be contraindicated due to P-gp interaction based upon data from the PALLAS trial. All patients will receive oral anticoagulation for stroke prevention according to current guideline recommendations.
  Interventions: Drug: Dronedarone
- Usual care (No Intervention): In most patients, the investigators anticipate usual care to include an atrioventricular nodal blocking agent (beta-blocker, non-dihydropyridine calcium channel blocker, or digoxin) without an antiarrhythmic. All patients will receive oral anticoagulation for stroke prevention according to current guideline recommendations.

INTERVENTIONS:
Drug: Dronedarone — Dronedarone 400 mg twice daily in addition to usual care
  Other Names: Multaq
  Arms: Dronedarone

SUMMARY:
While there are several completed clinical trials that address treatment strategy in patients with symptomatic and recurrent AF, there are no randomized clinical trials that address treatment for first-detected AF. In usual care, these patients are started on an atrioventricular nodal blocking agent (beta-blocker or non-dihydropyridine calcium channel blocker) along with stroke prevention therapy. The investigators hypothesize that earlier administration of a well-tolerated antiarrhythmic drug proven to reduce hospitalization may result in improved cardiovascular outcomes and quality of life in patients first-detected AF.

The purpose of this study is to determine if treatment with dronedarone on top of usual care is superior to usual care alone for the prevention of cardiovascular hospitalization or death from any cause in patients hospitalized with first-detected AF. All patients will be treated with guideline-recommended stroke prevention therapy according to the CHA2DS2-VASc score. The treatment follow-up period will be 12 months. There will be two follow-up visits. Consistent with the pragmatic nature of the trial, the first follow-up will occur between 3 -9 months and the 2nd will occur at 12 months (with a window of +/- 30 days). Approximately 3000 patients will be enrolled and randomly assigned (1:1) to study intervention. The study intervention will be dronedarone 400 mg twice daily in addition to usual care versus usual care alone.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia encountered in clinical practice, accounting for one-third of arrhythmia-related hospitalizations.1 As many as 1 in 4 people develop AF over their lifetime after the age of 40 years. The prevalence and burden of AF in the United States is substantial; the age-adjusted incidence and prevalence has increased over the last 3 decades. Moreover, the number of Americans with AF is expected to increase 150% by 2050. The goals of care in the treatment of AF include (1) the management and reduction of risk factors, (2) prevention of tachycardia (rate control), (3) prevention of stroke, and (4) improvement of symptoms. Reduction or elimination of symptoms often requires rhythm control. Historically, randomized clinical trials have not demonstrated a mortality or stroke benefit with a rhythm control versus a rate control strategy.

Despite the failure of prior randomized clinical trials to demonstrate the superiority of rhythm control, the recent Early Treatment of Atrial Fibrillation for Stroke Prevention 4 (EAST-AFNET 4) trial demonstrated that early introduction of a comprehensive rhythm-control strategy (within one year of diagnosis) is superior to guideline-based usual care in improving cardiovascular (CV) outcomes at a mean follow-up of 5 years. The EAST-AFNET 4 trial found that early rhythm control reduced the primary outcome of CV death, stroke, hospitalization for heart failure (HF), or acute coronary syndrome (HR 0.79, 96% confidence interval (CI) 0.66-0.94, p = 0.005). EAST-AFNET 4 also demonstrated a reduction in the risk of stroke with early introduction of rhythm control (HR 0.65, 95% CI 0.44-0.98), a finding that was also observed with dronedarone in the ATHENA trial. In addition, maintenance of sinus rhythm has been associated with improved quality of life and increased exercise capacity in some patients. Outside of clinical trials, a quality-of-life study from the Registry on Cardiac Rhythm Disorders Assessing the Control of Atrial Fibrillation (RECORD-AF) found that rhythm control was associated with better quality of life.

There are several antiarrhythmic drugs (AADs) available for rhythm control of AF. Class I antiarrhythmic agents are predominantly limited to younger patients without coronary artery or structural heart disease. Patients with advanced chronic kidney disease, prolonged QT intervals, and/or severe left ventricular hypertrophy should not be treated with sotalol or dofetilide. Even when sotalol or dofetilide can be used, patients are often hesitant to start a medication that requires an inpatient hospitalization for drug loading and laboratory evaluation every 3 months. Amiodarone has been shown to be the most effective AAD for maintaining sinus rhythm in patients with AF; however, based on its side effect profile, amiodarone is only recommended as a first-line agent under specific clinical circumstances. Moreover, despite its efficacy, amiodarone has high rates of discontinuation due to frequent adverse events. In addition to its unfavorable side effects, several studies, including those of patients at risk for sudden cardiac death, have demonstrated an association between amiodarone use and higher mortality, as well as lower functional status. In contrast to amiodarone, dronedarone is a much better tolerated antiarrhythmic medication. In randomized controlled trials, dronedarone has been shown to prevent recurrent AF, improve rate control, and decrease cardiovascular hospitalization in patients with AF.

While there are several completed clinical trials that address treatment strategy in patients with symptomatic and recurrent AF, there are no randomized clinical trials that address treatment for first-detected or new-onset AF. After appropriate evaluation for oral anticoagulation, these patients are often started on an atrioventricular nodal blocking agent (beta-blocker or non-dihydropyridine calcium channel blocker). The investigators hypothesize that earlier administration of a well-tolerated antiarrhythmic drug proven to reduce hospitalization may result in improved quality of life and cardiovascular outcomes in patients with first-detected AF.

Risk Assessment:

Dronedarone is approved by the Food and Drug Administration to reduce the risk of hospitalization for AF in patients with paroxysmal or persistent AF. The efficacy and safety of dronedarone 400 mg twice daily was evaluated in five controlled studies, ATHENA, ANDROMEDA, European Trial in Atrial Fibrillation or Flutter Patients Receiving Dronedarone for the Maintenance of Sinus Rhythm (EURIDIS), ADONIS, and Dronedarone Atrial FibrillatioN study after Electrical Cardioversion (DAFNE), involving more than 6,000 patients with including more than 3200 patients who received dronedarone. As with any therapeutic agent, there are known risks with dronedarone therapy. These risks include hepatic injury, heart failure exacerbation, increased exposure to digoxin, increased plasma concentration of tacrolimus, sirolimus, and other Cytochrome P450, family 3, subfamily A (CYP 3A) substrates, and very rare instances of pulmonary toxicity. The risks of dronedarone are felt to be outweighed by its benefits. The guideline recommendations provided by the European Society of Cardiology and American Heart Association (AHA)/American College of Cardiology (ACC)/Heart Rhythm Society (HRS) are commensurate with this risk benefit assessment.

Benefit Assessment:

While there are no completed randomized clinical trials to guide selection or initiation of rhythm control therapies in patients with first-detected AF, there are recent trials that suggest benefit with both dronedarone antiarrhythmic therapy and early-initiation of rhythm control in persons with AF. the recent EAST-AFNET 4 trial demonstrated that early introduction of a comprehensive rhythm-control strategy (within one year of diagnosis) is superior to usual guideline-recommended care in improving cardiovascular (CV) outcomes at 5 years. The median time from new-onset AF to randomization in the EAST-AFNET4 trial was 36 days. The trial found that early rhythm control reduced the primary outcome of CV death, stroke, hospitalization for HF, or acute coronary syndrome (HR 0.79, 95% confidence interval 0.66-0.94, p = 0.005). EAST-AFNET 4 also demonstrated a reduction in the risk of stroke with early introduction of rhythm control (HR 0.65, 95% CI 0.44-0.98), a finding that was also observed with dronedarone in the ATHENA trial. Thus, the investigators hypothesize that early initiation of dronedarone in patients with new-onset AF will lead to a reduction in CV hospitalization or death.

Overall Design:

Dronedarone is approved by the Food and Drug Administration to reduce the risk of CV hospitalization in patients with AF or atrial flutter. However, it is unknown if dronedarone (or any antiarrhythmic medication) can reduce CV hospitalization or death in patients with first-detected AF. This trial has been designed to address this important question. In order to facilitate the trial enrollment, data collection, and a generalizability to clinical practice, the CHANGE AFIB study has been designed as an open-label pragmatic clinical trial nested within the Get With The Guidelines (GWTG) Atrial Fibrillation registry. At present the overall GWTG program is being implemented in over 2,300 hospitals across the U.S. and is comprised of over 9 million patient records, with an estimated 650,000 new patient records entered per year. The trial will utilize the existing GWTG registry network, data collection architecture, and experience to facilitate both enrollment and conduct of the trial.

The comparator arm will be "usual care." Thus, this study will compare usual care plus dronedarone versus usual care alone. In most patients, the investigators anticipate usual care to include an atrioventricular nodal blocking agent (beta-blocker, non-dihydropyridine calcium channel blocker, or digoxin) without an antiarrhythmic. As dronedarone has anti-adrenergic rate controlling properties, a low dose of beta-blocker or calcium-channel blocker is recommended in the USPI when starting dronedarone. In the dronedarone arm concomitant digoxin use will be contraindicated due to P-gp interaction based upon data from the PALLAS trial. All patients will receive oral anticoagulation for stroke prevention according to current guideline recommendations.

CHANGE AFIB will leverage several critical advantages as a pragmatic clinical trial. Data collection will be integrated into the Get With The Guidelines AFIB registry. The use of the GWTG-AFIB registry will also enhance subject recruitment and ensure the enrollment of a diverse group of patients. The randomized intervention will be compared with usual care thus further enhancing generalizability. Follow-up visits will be minimized to reduce patient burden. Moreover, follow-up visits will have "windows" to accommodate variation in follow-up intervals at different centers.

Justification for Study Drug Intervention and Dose:

Dronedarone is a non-iodinated benzofuran similar to amiodarone but is not associated with thyroid or pulmonary toxicity in randomized clinical trials or post-marketing observational studies. Dronedarone has electrophysiological characteristics spanning all 4 Vaughan-Williams anti-arrhythmic classes, with primarily class III effects. Initial trials suggested that dronedarone prolonged the time to recurrence of AF and reduced cardiovascular death and hospitalization.

The landmark ATHENA trial evaluated the efficacy and safety of dronedarone in patients with atrial arrhythmias (atrial fibrillation or atrial flutter). This trial did not include patients with a recent history of New York Heart Association (NYHA) class IV heart failure or recent hospitalization for decompensated heart failure (<4 weeks). Approximately, 30% of the ATHENA population had NYHA class I-III heart failure. ATHENA demonstrated that dronedarone 400 mg twice daily (in combination with background therapy) reduced the combined endpoint of CV hospitalization or death from any cause by 24% (p<0.001) compared with placebo. Of course, the ATHENA trial was not conducted in the special population of patients with a new diagnosis of AF. There are no randomized trials or guideline recommendations for antiarrhythmic therapy at the time of first-detected AF. A subgroup analysis from the ATHENA trial suggests that optimal outcomes may be achieved in those patients with shorter duration of AF (time from diagnosis). Similar observations have also been made in patients undergoing other forms of rhythm control, including catheter ablation. In this trial, patients with first-detected AF will be randomized to dronedarone on top of usual care versus usual care alone. Patients randomized to the intervention arm will be prescribed and treated with Dronedarone 400 mg bid. This dose has been chosen as it is the Food and Drug Administration approved dose as well as the dose recommended in current international guidelines. Dronedarone has also been shown to be an effective rate control agent as well. In the ERATO study treatment with dronedarone 400 mg twice daily let to a mean reduction of 24.5 beat/min in patients with permanent AF when compared with placebo. In the EURIDIS/ADONIS studies the mean difference in patients with paroxysmal/persistent AF during AF recurrence was 14 beats/min. Moreover, the dronedarone treated patients experienced improved rate control without any reduction in exercise tolerance as measured by maximal exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=21 years.
2. First-detected atrial fibrillation (defined as atrial fibrillation diagnosed in the previous 120 days).
3. Electrocardiographic documentation of atrial fibrillation.
4. Estimated life expectancy of at least 1 year.
5. Patient or legal authorized representative capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Patients with prior or planned treatment with rhythm control, either catheter ablation or chronic (>7 days) antiarrhythmic drug therapy.

3. Planned cardiothoracic surgery. 4. New York Heart Association class III or IV heart failure or a hospitalization for heart failure in the last 4 weeks.

5. Patients with reduced ejection fraction (LVEF ≤40%). 6. Permanent atrial fibrillation. 7. Ineligible for oral anticoagulation, unless CHA2DS2-VASc is less than 3 in women or 2 in men.

8. Bradycardia with a resting heart rate < 50 bpm 9. PR interval >280 msec or 2nd degree or 3rd degree atrioventricular block without a permanent pacemaker/cardiac implanted electronic device.

10. Corrected QT interval >=500 msec. 11. Pregnancy or breast feeding. 12. Severe hepatic impairment in the opinion of the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Hospitalization or Death | Evaluated through 12 months from randomization
  First occurrence of unplanned CV hospitalization or death from any cause within 12 months of randomization. All unplanned hospitalizations (i.e. admission with an overnight stay in an acute care healthcare facility/hospital) for cardiovascular causes will be considered a cardiovascular hospitalization.

SECONDARY OUTCOMES:
Win Ratio | Evaluated through 12 months from randomization
  Among the randomized patients, every patient in the dronedarone arm will be compared with every patient in the usual care arm. Within each pair of patients, the component outcomes will be compared in descending order of importance until one of the patients in the pair demonstrates a better outcome compared with the other. For the purpose of this trial the hierarchy of component outcomes are shown below. The components in the WIN ratio hierarchy are similar to the endpoints considered in the recent EAST AFNET4 trial.
  Hierarchy of Outcomes for the WIN Ratio:
  1. All-cause mortality
  2. Ischemic stroke or systemic embolism
  3. Hospitalization for new/worsening diagnosis of heart failure
  4. Hospitalization for acute coronary syndrome
All-cause mortality | Evaluated through 12 months from randomization
  For descriptive purposes, deaths will be categorized by the site investigators according to the following categories: cardiovascular and non-cardiovascular. Cardiovascular deaths will be further classified into arrhythmic vs non-arrhythmic according the modified Hinkle-Thaler criteria, as used in several landmark cardiovascular trials. Patients who are well and (1) have a witnessed sudden collapse or (2) those found dead, but known to be alive and well in the previous 24 hours (e.g. no signs or symptoms of cardiorespiratory distress) will be defined as having arrhythmic death.
Ischemic stroke or systemic embolism | Evaluated through 12 months from randomization
  The occurrence of ischemic stroke will be defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction. Symptoms or signs must persist ≥24 hours, unless the stroke is documented by CT, MRI or autopsy, in which case the duration of symptoms/signs may be less than 24 hours. Stroke may be classified as ischemic (including hemorrhagic transformation of ischemic stroke), hemorrhagic, or undetermined. Systemic embolism will be defined as acute arterial insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g., trauma, atherosclerosis, or instrumentation).
Hospitalization for new/worsening diagnosis of heart failure | Evaluated through 12 months from randomization
  Hospitalization for new or worsening heart failure will be defined as any unplanned hospitalization (i.e. admission with an overnight stay in an acute care healthcare facility/hospital) due to a new diagnosis or worsening symptomatic heart failure
Hospitalization for acute coronary syndrome | Evaluated through 12 months from randomization
  Any hospitalization (i.e. admission with an overnight stay in an acute care healthcare facility/hospital) due to acute coronary syndrome.
Time to first unplanned cardiovascular hospitalization | Evaluated through 12 months from randomization
  Given the importance of CV hospitalization as an outcome from a clinical perspective, patient perspective, and economic perspective, there will be two analyses of CV hospitalization. The key secondary endpoint will be time to first unplanned CV hospitalization (similar to the component of the primary endpoint).
Unplanned cardiovascular hospitalizations--secondary analysis using Anderson-Gill extension | Evaluated through 12 months from randomization
  Given the importance of CV hospitalization as an outcome from a clinical perspective, patient perspective, and economic perspective, there will be two analyses of CV hospitalization. The second exploratory analysis of unplanned cardiovascular hospitalization will use a method to account for repeated events (Anderson-Gill extension).

OTHER OUTCOMES:
Any unplanned arrhythmia-related hospitalization | Evaluated through 12 months from randomization
  Arrhythmia-Related Hospitalization will be defined as any unplanned hospitalization (i.e. admission with an overnight stay in an acute care healthcare facility/hospital) due to any tachy or brady-arrhythmia.
Number of participants who experience AF progression | Evaluated through 12 months from randomization
  AF Progression will be defined as the transition from (a) paroxysmal to persistent or (b) persistent to permanent AF.
Number of participants who undergo cardioversion (pharmacologic or electrical) | Evaluated through 12 months from randomization
  Cardioversion (either pharmacologic or electrical) with or without transesophageal echocardiographic guidance will be a tertiary endpoint.
Number of participants who have ablation of AF (catheter, surgical or hybrid) performed | Evaluated through 12 months from randomization
  Ablation of AF including catheter ablation, surgical ablation, or hybrid (endocardial and epicardial ablation) ablation will be a tertiary endpoint.
Days alive and outside of the hospital | Evaluated through 12 months from randomization
  Days Alive and Out of the Hospital. Days alive and out of the hospital (DAOH, also referred to as "home time") is an emerging clinical trial endpoint that is both pragmatic and patient centered. It is highly correlated with traditional time-to-event mortality and hospitalization outcomes.
Patient-Reported Quality of Life--AFEQT | At baseline and 12 months
  The AFEQT is a 21-item, AF-specific health-related QOL questionnaire that assesses the impact of AF on patient-reported quality of life. The AFEQT includes a summary score (calculated from 18 of the questions) and subscale scores in three domains: symptoms, daily activities, and treatment concern. The summary and subscale scores range from 0 (corresponds to complete AF-related disability) to 100 (no AF-related disability). A change of 5 or more points in the AFEQT has been identified as a benchmark for a clinically meaningful difference in an individual patient.
Patient-Reported Quality of Life--MAFSI | At baseline and 12 months
  The MAFSI was developed as a modification and update of the AF Symptom Checklist. The trial will use a modified MAFSI questionnaire comprised of a 10-item AF symptom checklist that asks about frequency and severity of each symptom. Frequency of symptoms is recorded as 0 (never), 1 (rarely), 2 (sometimes), 3 (often), or 4 (always). These responses are summed for a total Frequency Score that ranges from 0 (no AF symptoms) to 40 (worst score). MAFSI Severity Scores are recorded as 1 (mild), 2 (moderate), or 3 (extreme). Severity scores are summed and range from 0 (no AF symptoms) to 30 (most severe AF symptoms). A clinically meaningful change in the MAFSI has not previously been established and therefore will be considered to be about ¼ of the pooled baseline standard deviation (SD), or 1.6 points for the Frequency Score and 1.3 points for the Severity Score.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Piccini, MD, MHS, Principal Investigator — Duke Clinical Research Organization
Locations (103):
- United States (103):
  - Thomas Hospital, Fairhope, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Los Angeles Medical Center (Kaiser Permenente), Los Angeles, California
  - West Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Medical Center (AKA UCI Health), Orange, California
  - Los Robles Health System - Los Robles Regional Medical Center, Thousand Oaks, California
  - UCLA Medical Center - Harbor, Torrance, California
  - Colorado Heart & Vascular Group - St. Anthony's Hospital, Lakewood, Colorado
  - Colorado Heart & Vascular Group - St. Anthony's North Health Campus, Westminster, Colorado
  - Christiana Hospital, Newark, Delaware
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Enmanuel Advanced Research Center, LLC, Miami, Florida
  - Life Spring Research Foundation, LLC, Miami, Florida
  - Nouvelle Clinical Research LLC, Miami, Florida
  - Golden Touch Clinical Research, Miami, Florida
  - Excellence Medical And Research, LLC, Miami, Florida
  - The Miami Research Group, Miami, Florida
  - Ocean Wellness Center, LLC, Miami Gardens, Florida
  - Pharma Medical Innovations, Miami Lakes, Florida
  - The Angel Medical Research, Miami Lakes, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Georgia Arrhythmia Consultants and Research Institute, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Mt Sinai Hospital Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - Riverside Medical Center, Kankakee, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Captain James A Lovell Federal Health Care Center, North Chicago, Illinois
  - Proctor Community Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Trinity Rock Island, Rock Island, Illinois
  - St. Elizabeth's Hospital of the Hospital Sisters of the Third Order of St. Francis, Springfield, Illinois
  - St. John's Hospital of the Hospital Sisters of the Third Order of St. Francis, Springfield, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Parkview Hospital, Inc., Fort Wayne, Indiana
  - Ascension St Vincent Hospital - Indianapolis, Indianapolis, Indiana
  - Kansas City Heart and Vascular Specialists at Providence Medical Center, Kansas City, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Adventist Healthcare Shady Grove Medical Center, Rockville, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - DMC Harper University Hospital (AKA Wayne State University Hospital), Detroit, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Trinity Health Ann Arbor Hospital - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - University Hospital - University of Missouri, Columbia, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Barnes-Jewish Hospital (AKA Washington Univ), St Louis, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - CHI Health Creighton University Medical Center - Bergan Mercy, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Albany Medical Center, Albany, New York
  - NewYork-Presbyterian/Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - NYC Health and Hospitals - Lincoln, The Bronx, New York
  - NYC Health and Hospitals - Jacobi, The Bronx, New York
  - NYC Health and Hospitals - North Central Bronx, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Durham VA Health Care System, Durham, North Carolina
  - WakeMed Raleigh Campus, Raleigh, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Trinity Hospital, Minot, North Dakota
  - The MetroHealth System, Cleveland, Ohio
  - Kettering Health Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - McLaren - St Lukes Hospital, Maumee, Ohio
  - Wooster Community Hospital Health System, Wooster, Ohio
  - Oklahoma City VA Health Care System, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Health Holy Spirit Medical Center, Camp Hill, Pennsylvania
  - Penn State Health Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Health St Joseph Medical Center - Main Campus, Reading, Pennsylvania
  - Ascension Saint Thomas Midtown, Nashville, Tennessee
  - Ascension Seton Medical Center Austin, Austin, Texas
  - Texas Health Fort Worth (FKA Texas Health Harris Methodist Hospital Fort Worth), Fort Worth, Texas
  - Memorial Hermann - Texas Medical Center, Houston, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Synapse Clinical Research, Missouri City, Texas
  - University Hospital at University of Texas San Antonio, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Chippenham and Johnston Willis Medical Center, Richmond, Virginia
  - Hunter Holmes McGuire VA Medical Center (AKA Richmond VA Medical Center), Richmond, Virginia
  - JW Ruby Memorial Hospital, Morgantown, West Virginia
  - Mayo Clinic Hospital - Franciscan Healthcare La Crosse, La Crosse, Wisconsin
  - UW Health at the American Center (AKA UW Health East Madison Hospital), Madison, Wisconsin
  - University Hospital - University of Wisconsin-Madison, Madison, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Medical Center, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wann LS, Curtis AB, January CT, Ellenbogen KA, Lowe JE, Estes NA 3rd, Page RL, Ezekowitz MD, Slotwiner DJ, Jackman WM, Stevenson WG, Tracy CM, Fuster V, Ryden LE, Cannom DS, Le Heuzey JY, Crijns HJ, Lowe JE, Curtis AB, Olsson SB, Ellenbogen KA, Prystowsky EN, Halperin JL, Tamargo JL, Kay GN, Wann LS, Jacobs AK, Anderson JL, Albert N, Hochman JS, Buller CE, Kushner FG, Creager MA, Ohman EM, Ettinger SM, Stevenson WG, Guyton RA, Tarkington LG, Halperin JL, Yancy CW; ACCF/AHA/HRS. 2011 ACCF/AHA/HRS focused update on the management of patients with atrial fibrillation (Updating the 2006 Guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2011 Jan 11;57(2):223-42. doi: 10.1016/j.jacc.2010.10.001. Epub 2010 Dec 21. No abstract available. PMID 21177058
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Feinberg WM, Blackshear JL, Laupacis A, Kronmal R, Hart RG. Prevalence, age distribution, and gender of patients with atrial fibrillation. Analysis and implications. Arch Intern Med. 1995 Mar 13;155(5):469-73. PMID 7864703
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Chamberlain AM, Gersh BJ, Alonso A, Chen LY, Berardi C, Manemann SM, Killian JM, Weston SA, Roger VL. Decade-long trends in atrial fibrillation incidence and survival: a community study. Am J Med. 2015 Mar;128(3):260-7.e1. doi: 10.1016/j.amjmed.2014.10.030. Epub 2014 Nov 8. PMID 25446299
- [Background] Novaro GM, Asher CR, Bhatt DL, Moliterno DJ, Harrington RA, Lincoff AM, Newby LK, Tcheng JE, Hsu AP, Pinski SL. Meta-analysis comparing reported frequency of atrial fibrillation after acute coronary syndromes in Asians versus whites. Am J Cardiol. 2008 Feb 15;101(4):506-9. doi: 10.1016/j.amjcard.2007.09.098. Epub 2007 Dec 20. PMID 18312767
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Furberg CD, Psaty BM, Manolio TA, Gardin JM, Smith VE, Rautaharju PM. Prevalence of atrial fibrillation in elderly subjects (the Cardiovascular Health Study). Am J Cardiol. 1994 Aug 1;74(3):236-41. doi: 10.1016/0002-9149(94)90363-8. PMID 8037127
- [Background] Psaty BM, Manolio TA, Kuller LH, Kronmal RA, Cushman M, Fried LP, White R, Furberg CD, Rautaharju PM. Incidence of and risk factors for atrial fibrillation in older adults. Circulation. 1997 Oct 7;96(7):2455-61. doi: 10.1161/01.cir.96.7.2455. PMID 9337224
- [Background] Benjamin EJ, Levy D, Vaziri SM, D'Agostino RB, Belanger AJ, Wolf PA. Independent risk factors for atrial fibrillation in a population-based cohort. The Framingham Heart Study. JAMA. 1994 Mar 16;271(11):840-4. PMID 8114238
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] Roy D, Talajic M, Nattel S, Wyse DG, Dorian P, Lee KL, Bourassa MG, Arnold JM, Buxton AE, Camm AJ, Connolly SJ, Dubuc M, Ducharme A, Guerra PG, Hohnloser SH, Lambert J, Le Heuzey JY, O'Hara G, Pedersen OD, Rouleau JL, Singh BN, Stevenson LW, Stevenson WG, Thibault B, Waldo AL; Atrial Fibrillation and Congestive Heart Failure Investigators. Rhythm control versus rate control for atrial fibrillation and heart failure. N Engl J Med. 2008 Jun 19;358(25):2667-77. doi: 10.1056/NEJMoa0708789. PMID 18565859
- [Background] Van Gelder IC, Hagens VE, Bosker HA, Kingma JH, Kamp O, Kingma T, Said SA, Darmanata JI, Timmermans AJ, Tijssen JG, Crijns HJ; Rate Control versus Electrical Cardioversion for Persistent Atrial Fibrillation Study Group. A comparison of rate control and rhythm control in patients with recurrent persistent atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1834-40. doi: 10.1056/NEJMoa021375. PMID 12466507
- [Background] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbuchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 1;383(14):1305-1316. doi: 10.1056/NEJMoa2019422. Epub 2020 Aug 29. PMID 32865375
- [Background] Ha AC, Breithardt G, Camm AJ, Crijns HJ, Fitzmaurice GM, Kowey PR, Le Heuzey JY, Naditch-Brule L, Prystowsky EN, Schwartz PJ, Torp-Pedersen C, Weintraub WS, Dorian P. Health-related quality of life in patients with atrial fibrillation treated with rhythm control versus rate control: insights from a prospective international registry (Registry on Cardiac Rhythm Disorders Assessing the Control of Atrial Fibrillation: RECORD-AF). Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):896-904. doi: 10.1161/HCQ.0000000000000011. Epub 2014 Nov 11. PMID 25387780
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Roy D, Talajic M, Dorian P, Connolly S, Eisenberg MJ, Green M, Kus T, Lambert J, Dubuc M, Gagne P, Nattel S, Thibault B. Amiodarone to prevent recurrence of atrial fibrillation. Canadian Trial of Atrial Fibrillation Investigators. N Engl J Med. 2000 Mar 30;342(13):913-20. doi: 10.1056/NEJM200003303421302. PMID 10738049
- [Background] Singh BN, Singh SN, Reda DJ, Tang XC, Lopez B, Harris CL, Fletcher RD, Sharma SC, Atwood JE, Jacobson AK, Lewis HD Jr, Raisch DW, Ezekowitz MD; Sotalol Amiodarone Atrial Fibrillation Efficacy Trial (SAFE-T) Investigators. Amiodarone versus sotalol for atrial fibrillation. N Engl J Med. 2005 May 5;352(18):1861-72. doi: 10.1056/NEJMoa041705. PMID 15872201
- [Background] AFFIRM First Antiarrhythmic Drug Substudy Investigators. Maintenance of sinus rhythm in patients with atrial fibrillation: an AFFIRM substudy of the first antiarrhythmic drug. J Am Coll Cardiol. 2003 Jul 2;42(1):20-9. doi: 10.1016/s0735-1097(03)00559-x. PMID 12849654
- [Background] Goldschlager N, Epstein AE, Naccarelli G, Olshansky B, Singh B. Practical guidelines for clinicians who treat patients with amiodarone. Practice Guidelines Subcommittee, North American Society of Pacing and Electrophysiology. Arch Intern Med. 2000 Jun 26;160(12):1741-8. doi: 10.1001/archinte.160.12.1741. PMID 10871966
- [Background] Packer DL, Prutkin JM, Hellkamp AS, Mitchell LB, Bernstein RC, Wood F, Boehmer JP, Carlson MD, Frantz RP, McNulty SE, Rogers JG, Anderson J, Johnson GW, Walsh MN, Poole JE, Mark DB, Lee KL, Bardy GH. Impact of implantable cardioverter-defibrillator, amiodarone, and placebo on the mode of death in stable patients with heart failure: analysis from the sudden cardiac death in heart failure trial. Circulation. 2009 Dec 1;120(22):2170-6. doi: 10.1161/CIRCULATIONAHA.109.853689. Epub 2009 Nov 16. PMID 19917887
- [Background] Fishbein DP, Hellkamp AS, Mark DB, Walsh MN, Poole JE, Anderson J, Johnson G, Lee KL, Bardy GH; SCD-HeFT Investigators. Use of the 6-min walk distance to identify variations in treatment benefits from implantable cardioverter-defibrillator and amiodarone: results from the SCD-HeFT (Sudden Cardiac Death in Heart Failure Trial). J Am Coll Cardiol. 2014 Jun 17;63(23):2560-2568. doi: 10.1016/j.jacc.2014.02.602. Epub 2014 Apr 9. PMID 24727258
- [Background] Thomas KL, Al-Khatib SM, Lokhnygina Y, Solomon SD, Kober L, McMurray JJ, Califf RM, Velazquez EJ. Amiodarone use after acute myocardial infarction complicated by heart failure and/or left ventricular dysfunction may be associated with excess mortality. Am Heart J. 2008 Jan;155(1):87-93. doi: 10.1016/j.ahj.2007.09.010. Epub 2007 Oct 25. PMID 18082495
- [Background] Saksena S, Slee A, Waldo AL, Freemantle N, Reynolds M, Rosenberg Y, Rathod S, Grant S, Thomas E, Wyse DG. Cardiovascular outcomes in the AFFIRM Trial (Atrial Fibrillation Follow-Up Investigation of Rhythm Management). An assessment of individual antiarrhythmic drug therapies compared with rate control with propensity score-matched analyses. J Am Coll Cardiol. 2011 Nov 1;58(19):1975-85. doi: 10.1016/j.jacc.2011.07.036. PMID 22032709
- [Background] Piccini JP, Hasselblad V, Peterson ED, Washam JB, Califf RM, Kong DF. Comparative efficacy of dronedarone and amiodarone for the maintenance of sinus rhythm in patients with atrial fibrillation. J Am Coll Cardiol. 2009 Sep 15;54(12):1089-95. doi: 10.1016/j.jacc.2009.04.085. PMID 19744618
- [Background] Hohnloser SH, Crijns HJ, van Eickels M, Gaudin C, Page RL, Torp-Pedersen C, Connolly SJ; ATHENA Investigators. Effect of dronedarone on cardiovascular events in atrial fibrillation. N Engl J Med. 2009 Feb 12;360(7):668-78. doi: 10.1056/NEJMoa0803778. PMID 19213680
- [Background] Singh BN, Connolly SJ, Crijns HJ, Roy D, Kowey PR, Capucci A, Radzik D, Aliot EM, Hohnloser SH; EURIDIS and ADONIS Investigators. Dronedarone for maintenance of sinus rhythm in atrial fibrillation or flutter. N Engl J Med. 2007 Sep 6;357(10):987-99. doi: 10.1056/NEJMoa054686. PMID 17804843
- [Background] Boriani G, Blomstrom-Lundqvist C, Hohnloser SH, Bergfeldt L, Botto GL, Capucci A, Lozano IF, Goette A, Israel CW, Merino JL, Camm AJ. Safety and efficacy of dronedarone from clinical trials to real-world evidence: implications for its use in atrial fibrillation. Europace. 2019 Dec 1;21(12):1764-1775. doi: 10.1093/europace/euz193. PMID 31324921
- [Background] Connolly SJ, Camm AJ, Halperin JL, Joyner C, Alings M, Amerena J, Atar D, Avezum A, Blomstrom P, Borggrefe M, Budaj A, Chen SA, Ching CK, Commerford P, Dans A, Davy JM, Delacretaz E, Di Pasquale G, Diaz R, Dorian P, Flaker G, Golitsyn S, Gonzalez-Hermosillo A, Granger CB, Heidbuchel H, Kautzner J, Kim JS, Lanas F, Lewis BS, Merino JL, Morillo C, Murin J, Narasimhan C, Paolasso E, Parkhomenko A, Peters NS, Sim KH, Stiles MK, Tanomsup S, Toivonen L, Tomcsanyi J, Torp-Pedersen C, Tse HF, Vardas P, Vinereanu D, Xavier D, Zhu J, Zhu JR, Baret-Cormel L, Weinling E, Staiger C, Yusuf S, Chrolavicius S, Afzal R, Hohnloser SH; PALLAS Investigators. Dronedarone in high-risk permanent atrial fibrillation. N Engl J Med. 2011 Dec 15;365(24):2268-76. doi: 10.1056/NEJMoa1109867. Epub 2011 Nov 14. PMID 22082198
- [Background] Kober L, Torp-Pedersen C, McMurray JJ, Gotzsche O, Levy S, Crijns H, Amlie J, Carlsen J; Dronedarone Study Group. Increased mortality after dronedarone therapy for severe heart failure. N Engl J Med. 2008 Jun 19;358(25):2678-87. doi: 10.1056/NEJMoa0800456. PMID 18565860
- [Background] Dagres N, Varounis C, Iliodromitis EK, Lekakis JP, Rallidis LS, Anastasiou-Nana M. Dronedarone and the incidence of stroke in patients with paroxysmal or persistent atrial fibrillation: a systematic review and meta-analysis of randomized trials. Am J Cardiovasc Drugs. 2011 Dec 1;11(6):395-400. doi: 10.2165/11594200-000000000-00000. PMID 22149318
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Hohnloser SH, Connolly SJ, Crijns HJ, Page RL, Seiz W, Torp-Petersen C. Rationale and design of ATHENA: A placebo-controlled, double-blind, parallel arm Trial to assess the efficacy of dronedarone 400 mg bid for the prevention of cardiovascular Hospitalization or death from any cause in patiENts with Atrial fibrillation/atrial flutter. J Cardiovasc Electrophysiol. 2008 Jan;19(1):69-73. doi: 10.1111/j.1540-8167.2007.01016.x. Epub 2007 Nov 21. PMID 18031520
- [Background] Ferreira JP, Jhund PS, Duarte K, Claggett BL, Solomon SD, Pocock S, Petrie MC, Zannad F, McMurray JJV. Use of the Win Ratio in Cardiovascular Trials. JACC Heart Fail. 2020 Jun;8(6):441-450. doi: 10.1016/j.jchf.2020.02.010. PMID 32466836
- [Background] Nieuwlaat R. The value of cardiovascular hospitalization as an endpoint for clinical atrial fibrillation research. Europace. 2011 May;13(5):601-2. doi: 10.1093/europace/eur119. No abstract available. PMID 21515593
- [Background] Amin AN, Jhaveri M, Lin J. Hospital readmissions in US atrial fibrillation patients: occurrence and costs. Am J Ther. 2013 Mar-Apr;20(2):143-50. doi: 10.1097/MJT.0b013e3182512c7e. PMID 23183097
- [Background] Hinkle LE Jr, Thaler HT. Clinical classification of cardiac deaths. Circulation. 1982 Mar;65(3):457-64. doi: 10.1161/01.cir.65.3.457. PMID 7055867
- [Background] Calkins H, Gliklich RE, Leavy MB, Piccini JP, Hsu JC, Mohanty S, Lewis W, Nazarian S, Turakhia MP. Harmonized outcome measures for use in atrial fibrillation patient registries and clinical practice: Endorsed by the Heart Rhythm Society Board of Trustees. Heart Rhythm. 2019 Jan;16(1):e3-e16. doi: 10.1016/j.hrthm.2018.09.021. Epub 2018 Nov 16. PMID 30449519
- [Background] Holmqvist F, Kim S, Steinberg BA, Reiffel JA, Mahaffey KW, Gersh BJ, Fonarow GC, Naccarelli GV, Chang P, Freeman JV, Kowey PR, Thomas L, Peterson ED, Piccini JP; ORBIT-AF Investigators. Heart rate is associated with progression of atrial fibrillation, independent of rhythm. Heart. 2015 Jun;101(11):894-9. doi: 10.1136/heartjnl-2014-307043. Epub 2015 Mar 2. PMID 25732748
- [Background] Fanaroff AC, Cyr D, Neely ML, Bakal J, White HD, Fox KAA, Armstrong PW, Lopes RD, Ohman EM, Roe MT. Days Alive and Out of Hospital: Exploring a Patient-Centered, Pragmatic Outcome in a Clinical Trial of Patients With Acute Coronary Syndromes. Circ Cardiovasc Qual Outcomes. 2018 Dec;11(12):e004755. doi: 10.1161/CIRCOUTCOMES.118.004755. PMID 30562068
- [Background] Greene SJ, O'Brien EC, Mentz RJ, Luo N, Hardy NC, Laskey WK, Heidenreich PA, Chang CL, Turner SJ, Yancy CW, Hernandez AF, Curtis LH, Peterson PN, Fonarow GC, Hammill BG. Home-Time After Discharge Among Patients Hospitalized With Heart Failure. J Am Coll Cardiol. 2018 Jun 12;71(23):2643-2652. doi: 10.1016/j.jacc.2018.03.517. PMID 29880124
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Calvert M, Kyte D, Mercieca-Bebber R, Slade A, Chan AW, King MT; the SPIRIT-PRO Group; Hunn A, Bottomley A, Regnault A, Chan AW, Ells C, O'Connor D, Revicki D, Patrick D, Altman D, Basch E, Velikova G, Price G, Draper H, Blazeby J, Scott J, Coast J, Norquist J, Brown J, Haywood K, Johnson LL, Campbell L, Frank L, von Hildebrand M, Brundage M, Palmer M, Kluetz P, Stephens R, Golub RM, Mitchell S, Groves T. Guidelines for Inclusion of Patient-Reported Outcomes in Clinical Trial Protocols: The SPIRIT-PRO Extension. JAMA. 2018 Feb 6;319(5):483-494. doi: 10.1001/jama.2017.21903. PMID 29411037
- [Background] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Holmes DN, Piccini JP, Allen LA, Fonarow GC, Gersh BJ, Kowey PR, O'Brien EC, Reiffel JA, Naccarelli GV, Ezekowitz MD, Chan PS, Singer DE, Spertus JA, Peterson ED, Thomas L. Defining Clinically Important Difference in the Atrial Fibrillation Effect on Quality-of-Life Score. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005358. doi: 10.1161/CIRCOUTCOMES.118.005358. PMID 31092022
- [Background] Packer DL, Piccini JP, Monahan KH, Al-Khalidi HR, Silverstein AP, Noseworthy PA, Poole JE, Bahnson TD, Lee KL, Mark DB; CABANA Investigators. Ablation Versus Drug Therapy for Atrial Fibrillation in Heart Failure: Results From the CABANA Trial. Circulation. 2021 Apr 6;143(14):1377-1390. doi: 10.1161/CIRCULATIONAHA.120.050991. Epub 2021 Feb 8. PMID 33554614
- [Background] Bubien RS, Knotts-Dolson SM, Plumb VJ, Kay GN. Effect of radiofrequency catheter ablation on health-related quality of life and activities of daily living in patients with recurrent arrhythmias. Circulation. 1996 Oct 1;94(7):1585-91. doi: 10.1161/01.cir.94.7.1585. PMID 8840848
- [Background] Wokhlu A, Monahan KH, Hodge DO, Asirvatham SJ, Friedman PA, Munger TM, Bradley DJ, Bluhm CM, Haroldson JM, Packer DL. Long-term quality of life after ablation of atrial fibrillation the impact of recurrence, symptom relief, and placebo effect. J Am Coll Cardiol. 2010 May 25;55(21):2308-16. doi: 10.1016/j.jacc.2010.01.040. PMID 20488300
- [Background] Hohnloser SH, Halperin JL, Camm AJ, Gao P, Radzik D, Connolly SJ; PALLAS investigators. Interaction between digoxin and dronedarone in the PALLAS trial. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1019-25. doi: 10.1161/CIRCEP.114.002046. Epub 2014 Nov 6. PMID 25378467
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Desai NR, Sciria CT, Zhao X, Piccini JP, Turakhia MP, Matsouaka R, Fonarow GC, Lewis WR. Patterns of Care for Atrial Fibrillation Before, During, and at Discharge From Hospitalization: From the Get With The Guidelines-Atrial Fibrillation Registry. Circ Arrhythm Electrophysiol. 2021 Apr;14(4):e009003. doi: 10.1161/CIRCEP.120.009003. Epub 2021 Mar 16. PMID 33724875
- [Background] Lewis WR, Piccini JP, Turakhia MP, Curtis AB, Fang M, Suter RE, Page RL 2nd, Fonarow GC. Get With The Guidelines AFIB: novel quality improvement registry for hospitalized patients with atrial fibrillation. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):770-7. doi: 10.1161/CIRCOUTCOMES.114.001263. Epub 2014 Sep 2. PMID 25185244
- [Background] Le Heuzey JY, De Ferrari GM, Radzik D, Santini M, Zhu J, Davy JM. A short-term, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of dronedarone versus amiodarone in patients with persistent atrial fibrillation: the DIONYSOS study. J Cardiovasc Electrophysiol. 2010 Jun 1;21(6):597-605. doi: 10.1111/j.1540-8167.2010.01764.x. Epub 2010 Apr 6. PMID 20384650
- [Background] Tave A, Goehring E, Desai V, Wu C, Bohn RL, Tamayo SG, Sicignano N, Juhaeri J, Jones JK, Weiss SR. Risk of interstitial lung disease in patients treated for atrial fibrillation with dronedarone versus other antiarrhythmics. Pharmacoepidemiol Drug Saf. 2021 Oct;30(10):1353-1359. doi: 10.1002/pds.5233. Epub 2021 May 4. PMID 33730412
- [Background] Blomstrom-Lundqvist C, Marrouche N, Connolly S, Corp Dit Genti V, Wieloch M, Koren A, Hohnloser SH. Efficacy and safety of dronedarone by atrial fibrillation history duration: Insights from the ATHENA study. Clin Cardiol. 2020 Dec;43(12):1469-1477. doi: 10.1002/clc.23463. Epub 2020 Oct 20. PMID 33080088
- [Background] Chew DS, Black-Maier E, Loring Z, Noseworthy PA, Packer DL, Exner DV, Mark DB, Piccini JP. Diagnosis-to-Ablation Time and Recurrence of Atrial Fibrillation Following Catheter Ablation: A Systematic Review and Meta-Analysis of Observational Studies. Circ Arrhythm Electrophysiol. 2020 Apr;13(4):e008128. doi: 10.1161/CIRCEP.119.008128. Epub 2020 Mar 19. PMID 32191539
- [Background] Davy JM, Herold M, Hoglund C, Timmermans A, Alings A, Radzik D, Van Kempen L; ERATO Study Investigators. Dronedarone for the control of ventricular rate in permanent atrial fibrillation: the Efficacy and safety of dRonedArone for the cOntrol of ventricular rate during atrial fibrillation (ERATO) study. Am Heart J. 2008 Sep;156(3):527.e1-9. doi: 10.1016/j.ahj.2008.06.010. PMID 18760136
- [Background] Gandhi SK, Reiffel JA, Boiron R, Wieloch M. Risk of Major Bleeding in Patients With Atrial Fibrillation Taking Dronedarone in Combination With a Direct Acting Oral Anticoagulant (From a U.S. Claims Database). Am J Cardiol. 2021 Nov 15;159:79-86. doi: 10.1016/j.amjcard.2021.08.015. PMID 34656316
- [Background] Xian Y, Fonarow GC, Reeves MJ, Webb LE, Blevins J, Demyanenko VS, Zhao X, Olson DM, Hernandez AF, Peterson ED, Schwamm LH, Smith EE. Data quality in the American Heart Association Get With The Guidelines-Stroke (GWTG-Stroke): results from a national data validation audit. Am Heart J. 2012 Mar;163(3):392-8, 398.e1. doi: 10.1016/j.ahj.2011.12.012. PMID 22424009
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Willi Maurer & Frank Bretz (2013) Multiple Testing in Group Sequential Trials Using Graphical Approaches, Statistics in Biopharmaceutical Research, 5:4, 311-320.
- [Background] Luo X, Tian H, Mohanty S, Tsai WY. An alternative approach to confidence interval estimation for the win ratio statistic. Biometrics. 2015 Mar;71(1):139-145. doi: 10.1111/biom.12225. Epub 2014 Aug 25. PMID 25156540
- [Background] Liu GF, Wang J, Liu K, Snavely DB. Confidence intervals for an exposure adjusted incidence rate difference with applications to clinical trials. Stat Med. 2006 Apr 30;25(8):1275-86. doi: 10.1002/sim.2335. PMID 16138360
- [Background] Jennison C and Turnbull BW. Group Sequential Methods with Applications to Clinical Trials. New York, NY: Chapman & Hall/CRC; 2000.
- [Derived] Pokorney SD, Nemeth H, Chiswell K, Albert C, Allyn N, Blanco R, Butler J, Calkins H, Elkind MSV, Fonarow GC, Fontaine JM, Frankel DS, Fermann GJ, Gale R, Kalscheur M, Kirchhof P, Koren A, Miller JB, Rashkin J, Russo AM, Rutan C, Steinberg BA, Piccini JP. Design and rationale of a pragmatic randomized clinical trial of early dronedarone versus usual care to change and improve outcomes in persons with first-detected atrial fibrillation - the CHANGE AFIB study. Am Heart J. 2025 Jan;279:66-75. doi: 10.1016/j.ahj.2024.10.001. Epub 2024 Oct 16. PMID 39423993